CLINICAL TRIAL: NCT02929888
Title: Effects of Intravenous Lysine Acetylsalicylate Versus Oral Aspirin on Platelet Responsiveness in Patients With ST-segment Elevation Myocardial Infarction: a Pharmacodynamic Study (ECCLIPSE-STEMI Trial)
Brief Title: Study of Platelet Function After Administration of Aspirin Versus Lysine Acetylsalicylate in STEMI Patients
Acronym: ECCLIPSE-STEMI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Responsible Party: Principal Investigator, David Vivas, MD, PhD, Fundacion Investigacion Interhospitalaria Cardiovascular
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-ECCLIPSESTEMI-01
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction
Keywords: ST-segment elevacion myocardial infarction, platelets
MeSH Terms: interventions — Aspirin

ARMS (2):
- Lysine Acetilsalicilate (LA) (Experimental): Loading dose (LD) of intravenous LA 450mg plus oral prasugrel 60mg/ticagrelor 180mg in patients with ST-segment elevation myocardial infarction
  Interventions: Drug: Lysine Acetilsalicilate
- Aspirin (Active Comparator): Loading dose (LD) of oral aspirin 300mg plus oral prasugrel 60mg/ticagrelor 180mg in patients with ST-segment elevation myocardial infarction
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Lysine Acetilsalicilate
  Arms: Lysine Acetilsalicilate (LA)
Drug: Aspirin
  Arms: Aspirin

SUMMARY:
Prasugrel and ticagrelor, new P2Y12-ADP receptor antagonists, are associated with greater pharmacodynamic inhibition and reduction of cardiovascular events in patients with an acute coronary syndrome. However, evidence is lacked about the effects of achieving faster and stronger cyclooxygenase inhibition with intravenous lysine acetylsalicylate (LA) compared to oral aspirin on prasugrel inhibited platelets. Recently, we demonstrated in healthy volunteers that the administration of intravenous LA resulted in a significantly reduction of platelet reactivity compared to oral aspirin on prasugrel inhibited platelets. Loading dose of LA achieves platelet inhibition faster, greater and with less variability than aspirin. However, there are no data of this issue in patients with an ST-segment elevation myocardial infarction (STEMI). The ECCLIPSE-STEMI trial will study the effect of LA versus aspirin in platelet reactivity in patients with STEMI

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center, open platelet function study conducted in 60 STEMI patients. Subjects were randomly assigned to receive a loading dose (LD) of intravenous LA 450mg plus oral prasugrel 60mg/ticagrelor 180mg, or LD of aspirin 300mg plus prasugrel 60mg/ticagrelor 180mg orally. Platelet function was evaluated at baseline, 30 min, 1h, 4h, and 24h using multiple electrode aggregometry and vasodilator-stimulated phosphoprotein phosphorylation (VASP). The primary endpoint of the study is the inhibition of platelet aggregation after arachidonic acid (AA) 1.5mM at 30 min. Secondary endopoints are the inhibition of platelet aggregation after AA baseline and at 1h, 4h and 24h, and measurement of aggregation with other platelet test (ADP, collagen and VASP).

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18.
* Patients with ST-segment myocardial infarction.
* Signed written informed consent.

Exclusion Criteria:

* Known allergies to aspirin, clopidogrel, prasugrel or ticagrelor.
* Cardiogenic shock or hemodinamic instability.
* Recent antiplatelet therapy (<14 days).
* Oral anticoagulation with a coumarin derivative.
* Any active bleeding or blood dyscrasia.
* Recent gastrointestinal bleeding (<6 months prior to inclusion).
* Recent history of stroke, TIA or intracranial bleeding (<6 months prior to inclusion).
* Known anemia, trombopenia or severe chronic kidney/liver disease
* Any known active neoplasm.
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation | 30 min
  The primary endpoint of the study, inhibition of platelet aggregation after arachidonic acid (AA) 1.5mM at 30 min

SECONDARY OUTCOMES:
Inhibition of platelet aggregation | 30 min, 1h, 4h, 24h
  Inhibition of platelet aggregation using different platelet function test (ADP, collagen, VASP)

CONTACTS AND LOCATIONS:
Overall Officials: David Vivas, MD, PhD, Principal Investigator — San Carlos University Hospital, Madrid, Spain
Locations (1):
- Fundacion, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Vivas D, Jimenez JJ, Martin-Asenjo R, Bernardo E, Ortega-Pozzi MA, Gomez-Polo JC, Moreno G, Vilacosta I, Perez-Villacastin J, Fernandez-Ortiz A. Effects of intravenous lysine acetylsalicylate versus oral aspirin on platelet responsiveness in patients with ST-segment elevation myocardial infarction: the ECCLIPSE-STEMI trial. J Thromb Thrombolysis. 2023 Feb;55(2):203-210. doi: 10.1007/s11239-022-02737-y. Epub 2022 Dec 8. PMID 36480147